CLINICAL TRIAL: NCT04124406
Title: Voyage: Real-World Impact of the Multi-target Stool DNA Test on CRC Screening and Mortality
Status: Active, not recruiting | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-08
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adults Prescribed Cologuard: Adults prescribed Cologuard for routine colon cancer screening by their healthcare provider.
  Interventions: Device: Cologuard

INTERVENTIONS:
Device: Cologuard — multi-target stool Deoxyribonucleic Acid (MT-sDNA) screening test

SUMMARY:
The purpose of this study is to gather information about the long term health of people who have been prescribed the Cologuard test, which is used for colorectal cancer (CRC) screening.

DETAILED DESCRIPTION:
Participates will be consented for prospective follow-up for health outcomes, which will be ascertained through periodic contacts. Participants will complete a baseline health questionnaire survey (T0) and a 1-year follow-up questionnaire survey (T1), allow access to medical records, when available, and allow future contacts for additional surveys.

ELIGIBILITY:
Inclusion Criteria:

* Resident of the United States
* Age 18 years or older
* Able to provide informed consent
* Able to complete surveys in English or Spanish
* Valid order for Cologuard screening

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults prescribed Cologuard for routine colon cancer screening by their healthcare provider.
Sampling Method: Probability Sample
Enrollment: 150000 (Estimated)
Dates: Start 2019-10-18 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Enrollment of Subjects | 3 years
  Enrollment of 150,000 subjects

SECONDARY OUTCOMES:
Diagnostic colonoscopy | 4.5 years
  Proportion having diagnostic colonoscopy within 1 year after positive CG test
CRC Frequency | 10 years
  Frequency of CRC among enrollees
National Rates Comparison | 10 years
  Comparison with national rates (i.e., SEER cancer registry rates) adjusted to reflect a) the age- and sex- distribution of CG users, b) that 25% of colorectal cancers occur in high risk patients, and c) the attrition rate of our longitudinal cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after de-identification. This may include text, tables, figures, and appendices. The study protocol (including statistical methods), informed consent form, and clinical study report will also be shared. Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available from 2 years and ending 4 years after publication.
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary IRB/EC approvals or waivers as applicable to conduct research.

REFERENCES:
- [Derived] Yost KJ, Carlson RE, Kirt CR, Kirsch EJ, Kneedler B, Laffin JJ, St Sauver JL, Finney Rutten LJ, Grimm JA, Olson JE. Recruitment strategies and consent rates in a national prospective colorectal cancer screening cohort: results from year 1 of the Voyage Study. BMJ Open Gastroenterol. 2024 Jul 17;11(1):e001376. doi: 10.1136/bmjgast-2024-001376. PMID 39019622
- [Derived] Olson JE, Kirsch EJ, Edwards V DK, Kirt CR, Kneedler B, Laffin JJ, Weaver AL, St Sauver JL, Yost KJ, Finney Rutten LJ. Colorectal cancer outcomes after screening with the multi-target stool DNA assay: protocol for a large-scale, prospective cohort study (the Voyage study). BMJ Open Gastroenterol. 2020 Feb 19;7(1):e000353. doi: 10.1136/bmjgast-2019-000353. eCollection 2020. PMID 32128228